CLINICAL TRIAL: NCT01773954
Title: Optical Coherence Tomography Guided Treat and Extend Therapy for Neovascular Age Related Macular Degeneration Using Aflibercept (the ATLAS Study)
Brief Title: Repeated Eye Injections of Aflibercept for Treatment of Wet Age Related Macular Degeneration
Acronym: ATLAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MidAtlantic Retina (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, MidAtlantic Retina, Investigator, Wills Eye
Organization: Wills Eye (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATLAS; 20122054 (Other: Western Institutional Review Board)
Record Dates: First submitted 2013-01-17; First posted 2013-01-23 (Estimated); Results first posted 2018-05-02 (Actual); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Age-Related Macular Degeneration; Macular Degeneration
Keywords: amd; age related macular degeneration; macular degeneration; neovascular
MeSH Terms: conditions — Macular Degeneration; Glycogen Storage Disease Type II

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intravitreal Aflibercept Injection More (Experimental): Patient receives treatment at baseline and week 4 visit. The first time extension criteria are met the follow-up interval will be increased by 4 weeks. Each time the extension criteria is met the interval will be extended by 2 weeks to a maximum of 16 weeks. If a patient is being followed at an 8 week interval but fails to meet extension criteria at a particular visit, treatment will be administered as usual and the follow up interval will be reduced to 4 weeks. If patient is being followed at 10-16 week interval but fails to meet extension criteria at a particular visit, treatment will be administered but the follow-up interval will be reduced by 2 week increments.
  Interventions: Drug: Intravitreal Aflibercept Injection

INTERVENTIONS:
Drug: Intravitreal Aflibercept Injection — Increased or decreased time between visits

SUMMARY:
To evaluate the visual outcome and number of injections required during an optical coherence tomography (OCT)-guided treat and extend regimen with intravitreal aflibercept for treatment of subfoveal neovascular age-related macular degeneration (NVAMD).

DETAILED DESCRIPTION:
The purpose of this study is to see how using "treat and extend," a method of determining how often a patient with NVAMD should visit the retina clinic and receive treatments, affects vision in patients with this condition after treatment. The treatment the investigators are using in this study is an eye injection of a drug called aflibercept (also called EYLEA). Eylea is FDA (Food and Drug Administration) approved for treatment of wet age related macular degeneration.

The investigators hope that "treat and extend" strikes the right balance between making sure patients get all of the treatments needed, but not giving patients too many treatments (so that the side effects of treatments are minimized and so that patients don't have to make more visits than they need to maintain maximum visual gain). The experimental part of this study is determining this "right balance" of eye injections.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 55 years with treatment naïve, active subfoveal NVAMD demonstrating macular fluid on optical coherence tomography (OCT) and leakage on fluorescein angiography (FA).
* Only one eye for each patient demonstrating a pre-treatment acuity of 20/25 - 20/320 is eligible
* Patients cannot have concurrent progressive retinal disease in the study eye.
* Willing and able to comply with clinic visits and study-related procedures
* Provide signed informed consent

Exclusion Criteria:

* Prior treatment for NVAMD in the study eye,
* Prior experimental treatment of NVAMD in either eye
* Prior treatment with systemic anti-VEGF (vascular endothelial growth factor) agents
* Prior treatment with verteporfin, plaque brachytherapy, or external-beam radiation therapy, or transpupillary thermotherapy in the study eye
* Previous subfoveal focal laser photocoagulation involving the foveal center in the study eye
* History of vitreo surgical intervention in the study eye. Cataract surgery is permitted.
* Concurrent eye disease in the study eye that could compromise visual acuity (e.g. diabetic retinopathy, advanced glaucoma)
* Any concurrent intraocular condition in the study eye (e.g. diabetic retinopathy or glaucoma) that, in the opinion of the investigator, could either
* require medical or surgical intervention during the 52 weeks study period to prevent or treat visual loss that might result from that condition, or
* allowed to progress untreated, could likely contribute to loss of at least 2 Snellen equivalent lines of best corrected visual acuity over the 52 weeks study period
* Active intraocular inflammation (grade trace or above) in the study eye, or history of idiopathic or autoimmune-associated uveitis in either eye
* Current vitreous hemorrhage in the study eye
* History of rhegmatogenous retinal detachment or macular hole (Stage 3 or 4) in the study eye
* Active infectious conjunctivitis, keratitis, scleritis, or endophthalmitis in either eye
* Aphakia, Anterior Chamber Intraocular Lens (ACIOL), or unstable Posterior Chamber Intraocular Lens (PCIOL).
* Uncontrolled glaucoma in the study eye (defined as intraocular pressure ≥30 mmHg despite treatment with anti-glaucoma medication)
* Pregnant or breast-feeding women
* Sexually active men* or women of childbearing potential** who are unwilling to practice adequate contraception during the study (adequate contraceptive measures include stable use of oral contraceptives or other prescription pharmaceutical contraceptives for 2 or more menstrual cycles prior to screening; intrauterine device [IUD]; bilateral tubal ligation; vasectomy; condom plus contraceptive sponge, foam, or jelly, or diaphragm plus contraceptive sponge, foam, or jelly)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carl Regillo, MD, Principal Investigator — Wills Eye Institute
Locations (3):
- United States (3):
  - Mid Atlantic Retina- Cherry Hill, Cherry Hill, New Jersey
  - Mid Atlantic Retina- Huntingdon Valley, Huntingdon Valley, Pennsylvania
  - Mid Atlantic Retina- Wills Eye Institute, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- Intravitreal Aflibercept: Intravitreal aflibercept on treat and extend schedule
Period: Overall Study
Arm/Group | Intravitreal Aflibercept
Started | 40
Completed | 31
Not Completed | 9

BASELINE CHARACTERISTICS:
Arm/Group | Intravitreal Aflibercept
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 81.3 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 17
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Best-corrected Early Treatment Diabetic Retinopathy Study (ETDRS) Letter Score
Time Frame: Baseline to Week 52
Measure: Mean (95% Confidence Interval); unit: letters
Arm/Group | Intravitreal Aflibercept
Number analyzed (Participants) | 40
letters | 7.2 [2.9 to 11.6]

2. Other Pre Specified Outcome: Change in Total Thickness at the Foveal Center Point on OCT
Time Frame: Baseline to Week 52
Measure: Mean (95% Confidence Interval); unit: micrometers
Arm/Group | Intravitreal Aflibercept
Number analyzed (Participants) | 40
micrometers | -143 [-187 to -99]

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Intravitreal Aflibercept
All-Cause Mortality (participants affected / at risk) | 2/40
Serious Adverse Events (participants affected / at risk) | 2/40
Other Adverse Events (participants affected / at risk) | 0/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intravitreal Aflibercept (N=40)
Fatal MI (Cardiac disorders) | 1
Endophthalmitis (Eye disorders) | 1

LIMITATIONS AND CAVEATS:
This is a non-controlled, non-comparative open label study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No